CLINICAL TRIAL: NCT04400474
Title: Exploratory Basket Trial of Cabozantinib Plus Atezolizumab in Advanced and Progressive Neoplasms of the Endocrine System. CABATEN Study
Brief Title: Trial of Cabozantinib Plus Atezolizumab in Advanced and Progressive Neoplasms of the Endocrine System. The CABATEN Study
Acronym: CABATEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: Ipsen (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETNE-T1914; 2019-002279-32 (EudraCT Number)
Record Dates: First submitted 2020-05-12; First posted 2020-05-22 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumor; Anaplastic Thyroid Cancer; Adenocarcinoma; Pheochromocytoma; Paraganglioma
Keywords: Cabozantinib; Atezolizumab
MeSH Terms: conditions — Neuroendocrine Tumors; Thyroid Carcinoma, Anaplastic; Adenocarcinoma; Pheochromocytoma; Paraganglioma | interventions — cabozantinib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib 40 mg + Atezolizumab 1200 mg (Experimental): * Cabozantinib 40 mg tablets, oral administration, once daily, continuously.
  * Atezolizumab 1200 mg administered intravenously, every three weeks (cycle).
  Interventions: Drug: Cabozantinib 40 mg

INTERVENTIONS:
Drug: Cabozantinib 40 mg — All the subjects will be treated with the combination of cabozantinib and atezolizumab until disease progression, unacceptable toxicity or patient consent withdrawal (whichever occurs first).
  Other Names: Atezolizumab 1200 mg

SUMMARY:
CABATEN is a multicohort phase II study of cabozantinib plus atezolizumab in advanced and progressive tumors from endocrine system.

The primary objective is to assess the efficacy of cabozantinib plus atezolizumab combination by means of radiological objective response rate (ORR) evaluated following RECIST v1.1 criteria in advanced endocrine tumors.

Endocrine tumors from different origins (thyroid, lung, pancreas and digestive tract, adrenal gland and paraganglia) are characterized by being remarkably vascular and expressing several growth factors including vascular endothelial growth factor (VEGF), platelet-derived growth factor (PDGF), insulin-like growth factor 1 (IGF-1), basic fibroblast growth factor (BFGF), and transforming growth factor (TGF)-α and -β. The (over) expression of some of these factors has been linked to poor prognosis. Cabozaninib, a VEGF inhibitor, in combination with atezolizumab, an inhibitor of PD-L1, may be active in endocrine tumors by overcoming the resistance to prior antiangiogenic drugs.

The trial will include patients with advanced and refractory tumors of endocrine system and patients would be allocated to six different cohorts according to the following tumor types.

DETAILED DESCRIPTION:
CABATEN is a multicohort phase II study of cabozantinib plus atezolizumab in advanced and progressive tumors from endocrine system.

Hypothesis:

The main hypothesis is that the administration of cabozantinib plus atezolizumab will improve the probability of expected objective response rate in advanced and refractory tumors of the endocrine system.

Objectives:

The primary objective is to assess the efficacy of cabozantinib plus atezolizumab combination by means of radiological objective response rate (ORR) evaluated following RECIST v1.1 criteria in advanced endocrine tumors. Secondary objectives include:

* To evaluate the safety profile of cabozantinib and atezolizumab combination, according to NCI-CTCAE V5.0.
* Duration of response (DoR) as per RECIST V1.1.
* Progression-free survival (PFS): median PFS as per RECIST V1.1.
* Overall Survival (OS): median OS as per RECIST V1.1.
* Tumor biomarkers: translational sub-study (optional).

Treatment:

All the subjects will be treated with the combination until disease progression, unacceptable toxicity, or patient consent withdrawal (whichever occurs first):

* Cabozantinib 40 mg or 20 mg tablets, oral administration once daily continuously.
* Atezolizumab 1200 mg administered intravenously (IV) every three weeks (cycle).

Rationale:

Endocrine tumors from different origins (thyroid, lung, pancreas and digestive tract, adrenal gland and paraganglia) are characterized by being remarkably vascular and expressing several growth factors including vascular endothelial growth factor (VEGF), platelet-derived growth factor (PDGF), insulin-like growth factor 1 (IGF-1), basic fibroblast growth factor (BFGF), and transforming growth factor (TGF)-α and -β. The (over) expression of some of these factors has been linked to poor prognosis. Cabozaninib, a VEGF inhibitor, in combination with atezolizumab, an inhibitor of PD-L1, may be active in endocrine tumors by overcoming the resistance to prior antiangiogenic drugs.

Patients allocation:

The trial will include patients with advanced and refractory tumors of endocrine system and patients would be allocated to six different cohorts according to the following tumor types:

Cohort 1: Well-differentiated neuroendocrine tumors of the lung and thymus (grades 1 and 2) after progression to somatostatin analogs, targeted agents, PRRT, and/or chemotherapy.

Cohort 2: Anaplastic thyroid cancer in first-line or after progression to chemotherapy or investigational drugs.

Cohort 3: Adrenocortical carcinoma after progression to chemotherapy and/or mitotane.

Cohort 4: Pheochromocytoma and paraganglioma after progression to peptide receptor radionuclide therapy (PRRT) if indicated, prior chemotherapy and biological therapy, such as somatostatin analogs, are allowed.

Cohort 5: Well-differentiated neuroendocrine tumors of digestive system after progression to somatostatin analogs, targeted agents, PRRT, and/or chemotherapy.

Cohort 6: Grade 3 neuroendocrine neoplasm of any origin, excluding small cell lung cancer, after progression to chemotherapy or targeted agents/PRRT.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 years old.
2. Willingness to participate in the study by signing informed consent form (ICF) approved by the trial Central Ethic Committee (CEIm).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Measurable disease per RECIST 1.1 as determined by the investigator.
5. Patients with an histopathologically confirmed disease (as per local pathology report), meeting one of the following (according to WHO 2010 classification):

   1. Cohort 1: Well-differentiated neuroendocrine tumours of the lung and thymus (WHO grade 1 and 2, typical and atypical carcinoids) after progression to somatostatin analogs, targeted agents, PRRT, and/or chemotherapy.
   2. Cohort 2: Anaplastic thyroid cancer in first-line or after progression to chemotherapy or investigational drugs. Primary tumour can be resected or not but risk of aerodigestive compression or bleeding should be ruled out.
   3. Cohort 3: Adrenocortical carcinoma after progression to chemotherapy and/or mitotane.
   4. Cohort 4: Pheochromocytoma and paraganglioma after progression to peptide receptor radionuclide therapy (PRRT) if indicated. Prior chemotherapy and biological therapy, such as somatostatin analogs, are allowed.
   5. Cohort 5: Well-differentiated neuroendocrine tumours of digestive system (WHO grade 1 and 2) after progression to somatostatin analogs, targeted agents, PRRT, and/or chemotherapy.
   6. Cohort 6: Grade 3 neuroendocrine neoplasm (WHO grade 3, including neuroendocrine (NET) and neuroendocrine carcinomas (NEC) G3) of any origin, excluding small cell lung cancer, after progression to chemotherapy or targeted agents/PRRT.
6. Recovery from toxicity related to any prior treatments to ≤ Grade 1, unless the adverse events (AEs) are clinically non-significant and/or stable on supportive therapy.
7. Ability to swallow tablets.
8. Adequate normal organ and marrow function as defined below:

   1. Haemoglobin ≥ 9.0 g/dL.
   2. Absolute neutrophil count (ANC) > 1500 per mm.
   3. Platelet count ≥ 100,000 per mm.
   4. Serum bilirubin ≤ 1.5x institutional upper limit of normal (ULN) unless liver metastases are present, in which case it must be ≤ 2X ULN. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology); however, they will be allowed only in consultation with their physician.
   5. Aspartate Transaminase (AST) (SGOT)/Alanine aminotransferase (ALT) (SGPT) ≤ 2.5x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 3x ULN.
   6. Measured creatinine clearance (CL) > 40 mL/min or Calculated creatinine CL > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for the determination of creatinine clearance.
9. Female subjects of childbearing potential (not surgically sterile or at least 2 years postmenopausal) must provide a negative urine pregnancy test at Screening, and use a medically accepted double barrier method of contraception (i.e condom with spermicide + IUD or cervical caps). In addition, they must agree to continue the use of this double barrier method for the duration of the study and for 4 months after participation in the study.
10. Males should agree to abstain from sexual intercourse with a female partner or agree to use a double barrier method of contraception (i.e.condom with spermicide, in addition to having their female partner use some contraceptive measures such as, intrauterine device (IUD) or cervical caps), for the duration of the study and for 4 months after participation in the study.
11. Willingness and ability of patients to comply with the protocol for the duration of the study including undergoing treatment as well as availability for scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Prior treatment with cabozantinib or any immune checkpoint inhibitor therapy (e.g, CTLA4, PD-1, or PD-L1 targeting agent).
2. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks or 5 half-lives of the agent, whichever is longer. Patients should have been out of mitotane for at least 4 weeks.
3. Receipt of any type of anticancer antibody (including investigational antibody) or systemic chemotherapy within 2 weeks before starting treatment.
4. Current or prior use of immunosuppressive medication within 2 weeks before the first dose of cabozantinib and atezolizumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
5. Active or prior documented autoimmune disease within the past 2 years. Note: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
6. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis).
7. History of allogeneic organ transplant.
8. Subjects having a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 28 days prior to the first dose of trial treatment.
9. Receipt of radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before inclusion. Subjects with clinically relevant ongoing complications from prior radiation therapy that have not completely resolved are not eligible (e.g, radiation esophagitis or other inflammation of the viscera).
10. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before inclusion. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of study treatment.
11. Concomitant anticoagulation with oral anticoagulants (e.g, warfarin, direct thrombin and factor Xa inhibitors) or platelet inhibitors (e.g, clopidogrel), except for the following allowed anticoagulants:

    * Low-dose aspirin for cardioprotection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
    * Anticoagulation with therapeutic doses of LMWH in subjects without known brain metastases and who are on a stable dose of LMWH for at least 6 weeks before inclusion and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumour.
12. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    a. Cardiovascular disorders: i. Class 3 or 4 congestive heart failure as defined by the New York Heart Association, unstable angina pectoris, and serious cardiac arrhythmias.

    ii. Uncontrolled hypertension defined as sustained blood press > 150 mm hg systolic or > 100 mm hg diastolic despite optimal antihypertensive treatment.

    iii. Stroke, including transient ischemic attack (TIA), myocardial infarction, other ischemic event, or thromboembolic event, e.g, deep venous thrombosis (DVT) and pulmonary embolism) within 6 months before inclusion. Subjects with a more recent diagnosis of DVT are allowed if stable, asymptomatic, and treated with LMWH for at least 6 weeks before study treatment.

    b. Gastrointestinal disorders (e.g, malabsorption syndrome or gastric outlet obstruction) including those associated with a high risk of perforation or fistula formulation: i. Tumours invading the GI tract, active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction. ii. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before inclusion. Note: complete healing of an intra-abdominal abscess must be confirmed prior to start of the treatment.

    c. Clinically significant hematemesis or hemoptysis of > 0.5 teaspoon (> 2.5 ml) of red blood or history of other significant bleeding within 3 months before treatment.

    d. Cavitating pulmonary lesion(s) or known endobronchial disease manifestation. e. Lesions invading major pulmonary blood vessels. f. Other clinically significant disorders such as: i. Active infection requiring systemic treatment, infection with human immunodeficiency virus or acquired immunodeficiency syndrome-related illness, or chronic hepatitis B or C infection.

    ii. Serious non-healing wound/ulcer/bone fracture. iii. Moderate to severe hepatic impairment (child-pugh B or C). iv. Requirement for hemodialysis or peritoneal dialysis. v. Uncontrolled diabetes mellitus. vi. History of solid organ transplantation.
13. Major surgery (e.g, GI surgery and removal or biopsy of brain metastasis) within 8 weeks before inclusion. Complete wound healing from major surgery must have occurred 4 weeks before study treatment and from minor surgery (e.g, simple excision, tooth extraction) at least 10 days before study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
14. Corrected QT interval calculated by the Fridericia formula (QTcf) > 500 ms within 28 days before study treatment.

    Note: if a single ECG shows a QTCf with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these 3 consecutive results for qtcf will be used to determine eligibility.
15. Pregnant or lactating females.
16. Inability to swallow tablets.
17. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
18. Diagnosis of another malignancy within 3 years before study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Capdevila, M.D, Ph.D, Study Chair — Hospital Universitari Vall d'Hebron, Barcelona
Locations (15):
- Spain (15):
  - Hospital Germans Trias i Pujol - ICO Badalona, Badalona, Barcelona
  - Hospital Duran i Reynals - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitario Elche, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LungNET (Lung Typical and Atypical Carcinoids): Lung typical and atypical carcinoids Cabozantinib 40 mg + Atezolizumab 1200 mg
- ATC (Anaplastic Thyroid Cancer): ATC in first-line or after PD to chemotherapy or investigational drugs Cabozantinib 40 mg + Atezolizumab 1200 mg
- ACC (Adrenocortical Carcinoma): ACC after PD to chemotherapy and/or mitotane Cabozantinib 40 mg + Atezolizumab 1200 mg
- PPGL (Pheochromocytoma/Paraganglioma): malignant PPGL (pheochromocytoma/paraganglioma) after PD to PRRT if indicated, prior chemotherapy and/or SSAs.
  Cabozantinib 40 mg + Atezolizumab 1200 mg
- G1-2 GEP-NET (Well-differentiated Gastroenteropancreatic NET): G1-2 GEP-NET, grade 1-2 gastroenteropancreatic NET Cabozantinib 40 mg + Atezolizumab 1200 mg
- G3 EP-NEN (Extrapulmonary Neuroendocrine Neoplasms.): G3 EP-NEN, grade 3 extrapulmonary neuroendocrine neoplasms. Cabozantinib 40 mg + Atezolizumab 1200 mg
Period: Overall Study
Arm/Group | LungNET (Lung Typical and Atypical Carcinoids) | ATC (Anaplastic Thyroid Cancer) | ACC (Adrenocortical Carcinoma) | PPGL (Pheochromocytoma/Paraganglioma) | G1-2 GEP-NET (Well-differentiated Gastroenteropancreatic NET) | G3 EP-NEN (Extrapulmonary Neuroendocrine Neoplasms.)
Started | 9 | 14 | 24 | 13 | 24 | 9
Completed | 9 | 14 | 24 | 13 | 24 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: patients with advanced and refractory endocrine and neuroendocrine neoplasms in 6 independent cohorts: well-differentiated neuroendocrine tumors (NET) of the lung (lungNET), anaplastic thyroid cancer (ATC), adrenocortical carcinoma (ACC), pheochromocytoma/paraganglioma (PPGL), well-differentiated gastroenteropancreatic NET (GEP-NET), and grade 3 extrapulmonary neuroendocrine neoplasms (G3 EP-NEN)
Groups:
- LungNET (Lung Typical Andatypical Carcinoids) Cabozantinib 40 mg + Atezolizumab 1200 mg: LungNET, Lung typical and atypical carcinoids Cabozantinib 40 mg + Atezolizumab 1200 mg
- ATC (Anaplastic Thyroid Cancer) Cabozantinib 40 mg + Atezolizumab 1200 mg: ATC in first-line or after PD to chemotherapy or investigational drugs Cabozantinib 40 mg + Atezolizumab 1200 mg
- ACC (Adrenocortical Carcinoma) Cabozantinib 40 mg + Atezolizumab 1200 mg: ACC after PD to chemotherapy and/or mitotane Cabozantinib 40 mg + Atezolizumab 1200 mg
- PPGL (Pheochromocytoma/Paraganglioma) Cabozantinib 40 mg + Atezolizumab 1200 mg: malignant PPGL (pheochromocytoma/paraganglioma) after PD to PRRT if indicated, prior chemotherapy and/or SSAs.
  Cabozantinib 40 mg + Atezolizumab 1200 mg
- Total: Total of all reporting groups
Arm/Group | LungNET (Lung Typical Andatypical Carcinoids) Cabozantinib 40 mg + Atezolizumab 1200 mg | ATC (Anaplastic Thyroid Cancer) Cabozantinib 40 mg + Atezolizumab 1200 mg | ACC (Adrenocortical Carcinoma) Cabozantinib 40 mg + Atezolizumab 1200 mg | PPGL (Pheochromocytoma/Paraganglioma) Cabozantinib 40 mg + Atezolizumab 1200 mg | G1-2 GEP-NET (Well-differentiated Gastroenteropancreatic NET) | G3 EP-NEN (Extrapulmonary Neuroendocrine Neoplasms.) | Total
Number analyzed (Participants) | 9 | 14 | 24 | 13 | 24 | 9 | 93
Age, Customized [Median (Full Range); unit: years]
  Age at inclusion | 63 [31 to 81] | 61.5 [47 to 80] | 50.5 [23 to 75] | 48.0 [36 to 67] | 59.5 [31 to 77] | 62.0 [38 to 73] | 59.0 [23 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 11 | 10 | 13 | 6 | 49
  Male | 5 | 9 | 13 | 3 | 11 | 3 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 9 | 14 | 24 | 12 | 23 | 9 | 91
  Race: Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race: African | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Radiological objective response rate (ORR) evaluated per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scan ORR= CR (confirmed complete response) + PR (confirmed partial response) as best response PR (At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: Through study completion, average 1 year
Population: Patients were enrolled in six cohorts. The main inclusion criteria were as follows: age > 18 years; Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0 or 1 and adequate organ and bone marrow function.
Measure: Count of Participants; unit: Participants
Groups:
- LungNET (Lung Typical Andatypical Carcinoids) Cabozantinib 40 mg + Atezolizumab 1200 mg: LungNET (Lung typical andatypical carcinoids) Cabozantinib 40 mg + Atezolizumab 1200 mg
Arm/Group | LungNET (Lung Typical Andatypical Carcinoids) Cabozantinib 40 mg + Atezolizumab 1200 mg | ATC (Anaplastic Thyroid Cancer) Cabozantinib 40 mg + Atezolizumab 1200 mg | ACC (Adrenocortical Carcinoma) Cabozantinib 40 mg + Atezolizumab 1200 mg | PPGL (Pheochromocytoma/Paraganglioma) Cabozantinib 40 mg + Atezolizumab 1200 mg | G1-2 GEP-NET (Well-differentiated Gastroenteropancreatic NET) | G3 EP-NEN (Extrapulmonary Neuroendocrine Neoplasms.)
Number analyzed (Participants) | 9 | 14 | 24 | 13 | 24 | 9
Participants | 0 | 2 | 2 | 2 | 4 | 0

2. Secondary Outcome: Safety Profile Number of Adverse Events Reactions (TRAEs)
Description: Number of patients adverse events reaction (TRAEs) related to Cabozantinib
Time Frame: TRAEs reported through clinical, up to 100 days after finishing or discontinuing treatment, on average 10 months
Population: Patients with advanced and refractory endocrine and neuroendocrine neoplasms, Patients were enrolled in six cohorts. The main inclusion criteria were as follows: age > 18 years; Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0 or 1 and adequate organ and bone marrow function
Measure: Count of Participants; unit: Participants
Arm/Group | LungNET (Lung Typical and Atypical Carcinoids) | ATC (Anaplastic Thyroid Cancer) | ACC (Adrenocortical Carcinoma) | PPGL (Pheochromocytoma/Paraganglioma) | G1-2 GEP-NET (Well-differentiated Gastroenteropancreatic NET) | G3 EP-NEN (Extrapulmonary Neuroendocrine Neoplasms.)
Number analyzed (Participants) | 9 | 14 | 24 | 13 | 24 | 9
Participants | 8 | 11 | 18 | 11 | 22 | 8

3. Secondary Outcome: Safety Profile Number of Adverse Events Reactions (TRAEs) Related With Atezolizumab
Description: Number of patients with adverse events reaction related to Atezolizumab as assessed by CTCAE v4.0
Time Frame: TRAEs reported through clinical, up to 100 days after finishing or discontinuing treatment, on average 10 months
Population: Patients with advanced and refractory endocrine and neuroendocrine neoplasms. Patients were enrolled in six cohorts. The main inclusion criteria were as follows: age > 18 years; Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0 or 1 and adequate organ and bone marrow function.
Measure: Count of Participants; unit: Participants
Arm/Group | LungNET (Lung Typical and Atypical Carcinoids) | ATC (Anaplastic Thyroid Cancer) | ACC (Adrenocortical Carcinoma) | PPGL (Pheochromocytoma/Paraganglioma) | G1-2 GEP-NET (Well-differentiated Gastroenteropancreatic NET) | G3 EP-NEN (Extrapulmonary Neuroendocrine Neoplasms.)
Number analyzed (Participants) | 9 | 14 | 24 | 13 | 24 | 9
Participants | 7 | 7 | 15 | 10 | 21 | 6

4. Secondary Outcome: Duration of Response (DoR)
Description: the time from the date of first documented CR or PR to the first documented progression or death due to underlying cancer. DoR will be determined based on tumour assessment (RECIST version 1.1 criteria).
Time Frame: From date of first documented clinical response (PR, CR) until the date of first documented progression, date of death from any cause or patient withdrawal, whichever came first, assessed up to 36 months
Population: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | ATC (Anaplastic Thyroid Cancer) | ACC (Adrenocortical Carcinoma) | PPGL (Pheochromocytoma/Paraganglioma) | G1-2 GEP-NET (Well-differentiated Gastroenteropancreatic NET)
Number analyzed (Participants) | 14 | 24 | 13 | 24
months | 20.4 [11.5 to 20.9] | 13.1 [5.4 to 20.9] | 12.2 [5.5 to 19.0] | 15.8 [10.6 to 20.2]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Median Progression free survival (mPFS) is defined as the time from the date of inclusion to the date of the first documented disease progression or death due to any cause, whichever occurs first. PFS will be determined based on tumour assessment (RECIST version 1.1 criteria). The local Investigator's assessments will be used for analyses.
Time Frame: From date of randomization until the date of first documented progression, date of death from any cause or patient withdrawal, whichever came first, assessed up to 36 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LungNET (Lung Typical and Atypical Carcinoids) | ATC (Anaplastic Thyroid Cancer) | ACC (Adrenocortical Carcinoma) | PPGL (Pheochromocytoma/Paraganglioma) | G1-2 GEP-NET (Well-differentiated Gastroenteropancreatic NET) | G3 EP-NEN (Extrapulmonary Neuroendocrine Neoplasms.)
Number analyzed (Participants) | 9 | 14 | 24 | 13 | 24 | 9
months | 8.4 [7.7 to NA] — 95% Confidence Interval is not reached due insufficient number of participants with events | 4.1 [2.7 to NA] — 95% Confidence Interval is not reached due insufficient number of participants with events | 2.9 [2.8 to 5.7] | 8.6 [5.7 to NA] — 95% Confidence Interval is not reached due insufficient number of participants with events | 13 [11.3 to NA] — 95% Confidence Interval is not reached due insufficient number of participants with events | 2.7 [2.6 to NA] — 95% Confidence Interval is not reached due insufficient number of participants with events

6. Secondary Outcome: Overall Survival (OS)
Description: Median Overall Survival (mOS) is calculated as the time from date of inclusion to date of death due to any cause.
Time Frame: Through study period, up to 3 years after completing treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LungNET (Lung Typical and Atypical Carcinoids) | ATC (Anaplastic Thyroid Cancer) | ACC (Adrenocortical Carcinoma) | PPGL (Pheochromocytoma/Paraganglioma) | G1-2 GEP-NET (Well-differentiated Gastroenteropancreatic NET) | G3 EP-NEN (Extrapulmonary Neuroendocrine Neoplasms.)
Number analyzed (Participants) | 9 | 14 | 24 | 13 | 24 | 9
months | NA [NA to NA] — not reached | 6.1 [4.4 to NA] — not reached | 13.5 [9.2 to NA] — not reached | 26.7 [9.7 to NA] — not reached | NA [NA to NA] — not reached | 5.4 [3.6 to NA] — not reached

ADVERSE EVENTS:
Time Frame: Adverse events will be reported through clinical study up to 100 days after the date of the decision to discontinue treatment, on average 3 years
Description: The SAE definition and reporting requirements are in accordance with the ICH Guideline for Clinical Safety Data Management: Definitions and Standards for Expedited Reporting, Topic E2A.
  The grade of adverse event will be coded according to the National Cancer Institute's Common Toxicity criteria (NCI-CTCAE v5.0 scoring system
Groups:
- Advanced and Refractory Endocrine and Neuroendocrine Neoplasms: Advanced and refractory endocrine and neuroendocrine neoplasms in 6 independent cohorts: well-differentiated neuroendocrine tumors (NET) of the lung (lungNET), anaplastic thyroid cancer (ATC), adrenocortical carcinoma (ACC), pheochromocytoma/paraganglioma (PPGL), well-differentiated gastroenteropancreatic NET (GEP-NET), and grade 3 extrapulmonary neuroendocrine neoplasms (G3 EP-NEN). All patients received atezolizumab 1200 mg IV Q3W plus cabozantinib 40 mg/day PO until disease progression or unacceptable toxicity.
  IMPORTANT: Adverse events were collected irrespective to the Arm/Group
Arm/Group | Advanced and Refractory Endocrine and Neuroendocrine Neoplasms
All-Cause Mortality (participants affected / at risk) | 2/93
Serious Adverse Events (participants affected / at risk) | 43/93
Other Adverse Events (participants affected / at risk) | 91/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced and Refractory Endocrine and Neuroendocrine Neoplasms (N=93)
Abdominal pain (Gastrointestinal disorders) | 7 (8)
Fever (General disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Alanine amino transferanse increased (Investigations) | 3 (3)
Aspatate amino ransferanse increased (Investigations) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
urinary tract infection (Endocrine disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
adrenal insufficiency (Endocrine disorders) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Lithiasis (Renal and urinary disorders) | 1 (1)
Covid-19 infection (Infections and infestations) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 1 (1) — Recto-vesical fistula infection
Small intestine infection (Infections and infestations) | 1 (1)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Tracheo-esophageal fistula
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
stroke (Nervous system disorders) | 1 (1) — ischemic stroke
Hemiplegia (Nervous system disorders) | 1 (1) — Left hemiplegia
Spinal cord compression surgery (Surgical and medical procedures) | 1 (1) — Spinal cord compression surgery
Brain metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Brain metastases. Treatment no-related secondary malignancy
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Infiltrating squamous cell carcinoma, moderately differentiated. No treatment related
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) — Acute cholangitis
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Inguinal pain
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Neoplasm related pain (acute and chronic)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced and Refractory Endocrine and Neuroendocrine Neoplasms (N=93)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 13 (23) — Gastrointestinal disorders - Other, specify
Abdominal pain (Gastrointestinal disorders) | 22 (26)
Infections and infestations - Other, specify (Infections and infestations) | 15 (18) — Infections and infestations - Other, specify
Fever (General disorders) | 12 (16)
General disorders and administration site conditions - Other, specify (General disorders) | 9 (10)
Diarrhea (Gastrointestinal disorders) | 44 (100)
Aspartate aminotransferase increased (Investigations) | 37 (82)
Alanine aminotransferase increased (Investigations) | 34 (81)
Vomiting (Gastrointestinal disorders) | 21 (41)
Constipation (Gastrointestinal disorders) | 13 (13)
Urinary tract infection (Infections and infestations) | 6 (8)
Fatigue (General disorders) | 67 (167)
Investigations - Other, specify (Investigations) | 22 (94)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 14 (18)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (15)
Edema limbs (General disorders) | 6 (7)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5)
Pain (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT04400474/Prot_SAP_000.pdf